CLINICAL TRIAL: NCT00470964
Title: Titanium-Sapphire Laser Trabeculoplasty in Glaucoma: A Randomized Study Comparing Titanium-Sapphire With Argon Laser Trabeculoplasty in Open-Angle Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goldschleger Eye Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 105-0011-001
Expanded Access: Available
Record Dates: First submitted 2007-05-06; First posted 2007-05-08 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Glaucoma, Open-Angle
Keywords: laser trabeculoplasty, glaucoma, argon, titanium-sapphire; IOP lowering effect; Adverse effects; IOP spikes
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Titanium Sapphire laser trabeculoplasty

SUMMARY:
Titanium Sapphire laser trabeculoplasty is effective in lowering intraocular pressure in glaucoma patients, and is comparable to argon laser trabeculoplasty

DETAILED DESCRIPTION:
Objective: To compare the medium-term outcome of Titanium-Sapphire laser trabeculoplasty (TiSLT) vs. Argon Laser Trabeculoplasty (ALT) in uncontrolled Open-angle Glaucoma (OAG) patients.

Methods: Prospective, masked, randomized comparative clinical study. Thirty-seven OAG patients with uncontrolled IOP and no previous filtration surgery (22 females and 15 males, mean age of 68 years) participated. Eighteen were treated with TiSLT and 19 with ALT. All patients underwent a comprehensive eye examination including visual acuity, IOP, goniocscopy and slit-lamp biomicroscopy and visual field examinations. Patients were examined pre-operatively and then at 1 hour, 1 day, 1 week, 1, 3 and 6 months, 1 year and 18 months post-operatively.

Main outcome measures: Final IOP, delta IOP and number of anti-glaucoma medications.

Results: The 18 patients in the TiSLT arm had an average of 8.3(±2.7) mm Hg or 32% reduction from pre-operative IOP (P<0.001). The 19 patients in the ALT arm had a mean IOP decrease of 6.5 (±4.3) mm Hg (P<0.001) or a 25% IOP reduction. Patients in both groups achieved a similar decrease in IOP (P>0.05). TiSLT patients had statistically significant fewer IOP spikes compared to the ALT group. (P=0.002). Two patients (1 in each arm) underwent trabeculectomy and were considered failures. Mean follow-up time was 15 months.

Conclusions: TiSLT provides similar efficacy to ALT in IOP reduction in OAG patients, and may offer better safety with fewer IOP spikes see post-operatively.

Application to clinical practice: If confirmed in additional studies, TiSLT may be used as an alternative to ALT in OAG patients.

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled open angle glaucoma patients

Ages: 40 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
IOP

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melamed, MD, Principal Investigator — Goldschleger Eye Institute
Locations (1):
- Goldschleger Eye Institute, Ramat Gan, Israel